CLINICAL TRIAL: NCT01032746
Title: Use of a Personal Health Record to Improve Colorectal Cancer Screening
Brief Title: Personal Electronic Health Records in Improving Screening Rates for Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Ayanian, Harvard Medical School
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Screening
Other Study IDs: CDR0000661288; HMS-11960
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Early Intervention, Educational; Occult Blood

INTERVENTIONS:
Other: educational intervention
Other: internet-based intervention
Procedure: evaluation of cancer risk factors
Procedure: fecal occult blood test
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Use of a web-based risk assessment tool may help improve screening rates for colorectal cancer.

PURPOSE: This randomized clinical trial is studying personal electronic health records to see how well they work in improving screening rates for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess whether screening rates for colorectal cancer (CRC) can be substantially increased among adults in primary care through the use of a personal electronic health record that provides a link to a validated web-based tool to estimate an individual's risk of CRC and electronic scheduling of CRC screening exams.

OUTLINE: This is a multicenter study. Participants are stratified according to participating Harvard Vanguard Medical Associates (HVMA) center. Participants are randomized to 1 of 2 arms.

* Intervention arm: Participants receive an electronic message within their MyHealth account on behalf of their primary care physician providing a link to a web-based tool to allow them to assess their personal risk of colorectal cancer (CRC). The tool provides an estimate of an individual's personal risk of developing different types of cancer over the next 10 years relative to others of the same age and sex. The tool also recommends steps that individuals can take to reduce their risk. The tool includes questions about family history; prior screening tests; dietary habits (red meat, fruits, and vegetables); weight and height; and use of folate, aspirin, estrogen therapy, alcohol, and tobacco. In addition, the electronic message provides information regarding options for CRC screening, emphasizing colonoscopy every 10 years per the current HVMA guidelines, followed by the secondary recommendation of annual fecal occult blood testing. Detailed information is provided in the form of a link to online educational materials. Participants may request either colonoscopy or fecal occult blood testing by responding to the electronic message and indicating their preference. Participants who request colonoscopy are contacted by the gastroenterology department to proceed with CRC screening; participants who request fecal occult blood testing will receive a stool card test kit in the mail from their primary care physician.
* Control arm: Participants receive no intervention.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Overdue for colorectal cancer screening (identified using automated extracts from the electronic medical record), as defined by the following criteria:

  * No fecal occult blood test within the past 12 months
  * No flexible sigmoidoscopy within the past 5 years
  * No colonoscopy within the past 10 years
* Receiving primary care at a Harvard Vanguard Medical Associates (HVMA) center
* Registered to use the HVMA patient portal (MyHealth) AND has an active MyHealth account

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-03; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Receipt of colorectal cancer screening exam (fecal occult blood test, flexible sigmoidoscopy, or colonoscopy) within 4 months following delivery of an electronic message within the personal health record

SECONDARY OUTCOMES:
Proportion of participants who access the web-based risk-assessment tool
Distribution of risk-status among participants who complete the web-based risk-assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: John Ayanian, MD, MPP, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Harvard Medical School, Boston, Massachusetts
  - Harvard Vanguard Medical Associates - Kenmore, Boston, Massachusetts

REFERENCES:
- [Result] Sequist TD, Zaslavsky AM, Colditz GA, Ayanian JZ. Electronic patient messages to promote colorectal cancer screening: a randomized controlled trial. Arch Intern Med. 2011 Apr 11;171(7):636-41. doi: 10.1001/archinternmed.2010.467. Epub 2010 Dec 13. PMID 21149743